CLINICAL TRIAL: NCT03909386
Title: Multicenter, Non-interventional Study on Patients With Atrial Fibrillation (AF) and Cancer (Diagnosed Within the Last 3 Years Prior to Enrolment)
Brief Title: Non-interventional Study on Patients With Atrial Fibrillation and Cancer
Acronym: BLITZ-AFCancer
Status: Completed | Type: Observational
Sponsor: Heart Care Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: K21
Record Dates: First submitted 2019-04-05; First posted 2019-04-10 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Atrial Fibrillation; Cancer
MeSH Terms: conditions — Atrial Fibrillation; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
AF and cancer frequently coexist. Since these patients are usually excluded from randomized trials, information on their management and outcome is scarce. Occurrence of relevant clinical events, such as ischemic and hemorrhagic and all-cause mortality and cardiovascular (CV) mortality occurring in patients treated or not with antithrombotic agents needs to be clarified.

A prospective observational registry collecting information, in a real world setting, on the clinical profile of patients with these clinical conditions and on the use of antithrombotic drugs in patients with AF and cancer could improve our knowledge on the management of these high risk patients.

DETAILED DESCRIPTION:
International, multicenter, non-interventional study on patients with atrial fibrillation (AF) and cancer (diagnosed within the last 3 years prior to enrolment).

The study will be conducted in about 80 sites in italy and 50 sites distributed in other European countries (Belgium, Germany, Ireland, Portugal, Spain, The Netherlands, Turkey).

The study will continue till the consecutive recruitment of 1500 patients. The recruitment period will last approximately 24 months.

Number of visits per patient: Baseline and 1 year (Final). Physicians will not be required to perform any additional tests, assessments, etc., not in line with their routine medical practice.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Age >18 years
* Patient with diagnosed AF (any type of AF, electrocardiographically documented within 1 year prior to enrolment)
* Patient with a documented cancer (diagnosed within the last 3 years prior to enrolment into this registry), including melanoma but not other basal-cell or squamous-cell carcinoma of the skin. The diagnosis/history of cancer must be objectively documented.
* Written informed consent (IC) for participation in the study
* Patient not simultaneously participating in any interventional study.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with diagnosed AF (any type of AF, electrocardiographically documented within 1 year prior to enrolment) and with a documented cancer (diagnosed within the last 3 years prior to enrolment into this registry), including melanoma but not other basal-cell or squamous-cell carcinoma of the skin. The diagnosis/history of cancer must be objectively documented.
Sampling Method: Non-Probability Sample
Enrollment: 1514 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Patients with AF and cancer treated with oral anticoagulant therapy and with other antithrombotic therapy | Baseline
  Number of patients with AF and cancer treated with oral anticoagulant therapy and with other antithrombotic therapy
Patients with AF and cancer treated with oral anticoagulant therapy and with other antithrombotic therapy | 12 Months
  Number of patients with AF and cancer treated with oral anticoagulant therapy and with other antithrombotic therapy

SECONDARY OUTCOMES:
Patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing all cause stroke | Baseline and 12 months
  Number of patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing all cause stroke
Patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing transient ischemic attacks | Baseline and 12 months
  Number of patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing transient ischemic attacks
Patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing major adverse cardiovascular events (non fatal MI, non fatal stroke, non fatal systemic embolic events, cardiovascular death) | Baseline and 12 months
  Number of patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing major adverse cardiovascular events (non fatal MI, non fatal stroke, non fatal systemic embolic events, cardiovascular death)
Patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing systemic embolic events | Baseline and 12 months
  Number of patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing systemic embolic events
Patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing acute coronary syndrome | Baseline and 12 months
  Number of patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing acute coronary syndrome
Patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing venous thromboembolic events, defined as composite of deep vein thrombosis and pulmonary embolism | Baseline and 12 months
  Number of patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing venous thromboembolic events, defined as composite of deep vein thrombosis and pulmonary embolism
Patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing deep vein thrombosis | Baseline and 12 months
  Number of patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing deep vein thrombosis
Patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing pulmonary embolism | Baseline and 12 months
  Number of patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing pulmonary embolism
Patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing major bleeding (Fatal bleeding, Non-fatal bleeding,Intracranial hemorrhage | Baseline and 12 months
  Number of patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing major bleeding (Fatal bleeding, Non-fatal bleeding,Intracranial hemorrhage
Patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing clinically relevant non-major bleeding | Baseline and 12 months
  Number of patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing clinically relevant non-major bleeding
Patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing composite of major and CRNM bleeding | Baseline and 12 months
  Number of patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing composite of major and CRNM bleeding
Patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing all-cause death | Baseline and 12 months
  Number of patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing all-cause death
Patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing cardiovascular death | Baseline and 12 months
  Number of patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing cardiovascular death
Patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing death due to malignancy | Baseline and 12 months
  Number of patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing death due to malignancy
Patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing sudden and unexplained death | Baseline and 12 months
  Number of patients treated with oral anticoagulant therapy, other antithrombotic therapy or not treated experiencing sudden and unexplained death
Association of various antithrombotic treatments (or lack of) on hospital admissions due to CV or non CV causes | Baseline and 12 months
  Number of hospital admissions (defined as ≥ 24 h stay in a hospital) due to CV or non CV causes
Association of various antithrombotic treatments (or lack of) on hospital admissions due to CV or non CV causes | Baseline and 12 months
  Length of hospital admissions (defined as ≥ 24 h stay in a hospital) due to CV or non CV causes;
Treatment satisfaction | Baseline and 12 months
  Treatment satisfaction as assessed by the Perception Anticoagulant Treatment Questionnaire (PACT-Q)
Quality of life satisfaction | Baseline and 12 months
  Health related quality of life as assessed by the EuroQol (EQ-5D-5L) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michele M Gulizia, MD, Study Chair — Heart Care Foundation
Locations (147):
- Belgium (12):
  - OLV ZIEKENHUIS AALST - Cardiology, Aalst
  - AZ IMELDA - Cardiology, Bonheiden
  - AZ ST-JAN - Cardiology, Bruges
  - Hôpital Erasme - Cardiology, Brussels
  - UCL Cliniques universitaires Saint-Luc - Cardiolgy, Brussels
  - UZ Brussel - Cardiology, Brussels
  - Ziekenhuis Oost-Limburg - Cardiology, Genk
  - JESSA HASSELT - Cardiology, Hasselt
  - AZ GROENINGE - Cardiology, Kortrijk
  - UZ LEUVEN - Cardiovascular diseases, Leuven
  - AZ DELTA ROESELARE - Cardiology, Roeselare
  - AZ TURNHOUT - Cardiology, Turnhout
- Ireland (3):
  - Bon Secours Hospital Cork - Oncology Department, Cork
  - Beacon Hospital, Cardiology, Dublin
  - Tallaght University Hospital - Geriatric and Stroke Medicine Department, Dublin
- Italy (100):
  - Ospedale San Giovanni Di Dio - Uo Cardiologia E Utic, Agrigento, AG
  - Ospedale Barone Lombardo - Cardiologia E Utic, Canicattì, AG
  - Ospedale Santo Spirito - Sc Cardiologia, Casale Monferrato, AL
  - Ospedale Civile Profili - U.O. Cardiologia, Fabriano, AN
  - Ospedale San Donato - U.O. Cardiologia, Arezzo, AR
  - Ospedale San Paolo - Cardiologia-Utic, Bari, BA
  - Istituto Tumori Giovanni Paolo Ii - U.O. Di Cardiologia, Bari, BA
  - Ospedali Treviglio-Caravaggio - Cardiologia, Treviglio, BG
  - Ospedale Civile - Sc Cardiologia, Belluno, BL
  - Ospedale Santa Maria Del Prato - U.O. Di Cardiologia, Feltre, BL
  - Ospedale Maggiore - U.O. Di Cardiologia, Bologna, BO
  - Ospedale Policlinico S. Orsola-Malpighi - U.O. Cardiologia-Rapezzi, Bologna, BO
  - Ospedale Bellaria - U.O. Di Cardiologia, Bologna, BO
  - Ospedale A. Businco - Servizio Di Cardiologia, Cagliari, CA
  - Ospedale Roberto Binaghi - Servizio Di Cardiologia, Cagliari, CA
  - Az. Ospedaliera S. Anna E S. Sebastiano - Cardiologia Clinica Universitaria - Utic, Caserta, CE
  - Ospedale San Giuseppe E Melorio - U.O.C. Cardiologia Utic, Santa Maria Capua Vetere, CE
  - Ospedale Regina Montis Regalis - U.O. Cardiologia-Utic, Mondovì, CN
  - Ospedale Maggiore Ss. Annunziata - Sc Cardiologia, Savigliano, CN
  - Ospedale Civile Ferrari - U.O.C. Cardiologia-Utic, Castrovillari, CS
  - Ospedale Spoke Paola- Cetraro Po Paola - Utic Cardiologia, Paola, CS
  - P.O. Garibaldi-Nesima - U.O.C. Di Cardiologia, Catania, CT
  - Azienda Ospedaliera Cannizzaro - Uoc Cardiologia Con Utic Ed Emodinamica, Catania, CT
  - Humanitas Centro Catanese Di Oncologia - Servizio Di Cardiologia, Catania, CT
  - Ospedali Riuniti - S.C. Di Cardiologia Univ.-Utic, Foggia, FG
  - Ospedale Civile San Giuseppe - Cardiologia, Empoli, FI
  - Ospedale San Giovanni Di Dio - Cardiologia, Florence, FI
  - Aou Careggi - Cardiologa Diagnostica, Florence, FI
  - Aou Careggi - Diagnostica Cardiovascolare, Florence, FI
  - Ospedale Policlinico San Martino - Clinica Malattie Cardiovascolari, Genova, GE
  - Ospedale Padre Antero Micone - Sc Cardiologia - Utic, Genova, GE
  - Ospedale San Giuseppe Da Copertino - U.O. Di Cardiologia-Utic, Copertino, LE
  - Ospedale Ignazio Veris Delli Ponti - Uoc Cardiologia-Utic, Scorrano, LE
  - Nuovo Ospedale Versilia - Sc Cardiologia, Lido di Camaiore, LU
  - Policlinico G. Martino - U.O. Medicina Interna, Messina, ME
  - Istituto Nazionale Tumori - Struttura Complessa Di Cardiologia, Milan, MI
  - Istituto Europeo Di Oncologia - Cardiologia, Milan, MI
  - Asst Ospedale Metropolitano Niguarda - Cardiologia 4 -Diagnost. E Riabilitativa, Milan, MI
  - Ospedale Di Vizzolo Predabissi - Uo Cardiologia E Ucc, Vizzolo Predabissi, MI
  - Ospedale Ramazzini - U.O. Cardiologia, Carpi, MO
  - Ospedale Di Sassuolo - Cardiologia, Sassuolo, MO
  - Ospedale San Francesco - Cardiologia - Utic, Nuoro, NU
  - Fondazione G. Giglio - U.O. Cardiologia E Utic, Cefalù, PA
  - Aor Villa Sofia-Cervello P.O. Cervello, Uo Cardiologia - Cervello, Palermo, PA
  - Istituto Oncologico Veneto - Cardiologia Oncologica, Padua, PD
  - Ospedale Civile Dello Spirito Santo - Utic E Cardiologia Interventistica, Pescara, PE
  - Azienda Ospedaliera Universitaria Pisana - U.O. Malattie Cardiovasc. I - Cisanello, Pisa, PI
  - Centro Di Riferimento Oncologico (Cro) - Cardiologia, Aviano, PN
  - Presidio Ospedaliero San Salvatore - Cardiologia E Utic, Pesaro, PU
  - Fondazione Irccs Policlinico San Matteo - Cardiologia, Pavia, PV
  - Ics Maugeri Spa Societa' Benefit - U.O. Di Riabilitazione Cardiologica, Pavia, PV
  - Ospedale Civile Santa Maria Delle Croci - U.O. Di Cardiologia, Ravenna, RA
  - Ospedale Santa Maria Degli Ungheresi - Uoc Cardiologia-Utic, Polistena, RC
  - Grande Ospedale Metropolitano-Bianchi Melacrino Morelli - Divisione Di Cardiologia, Reggio Calabria, RC
  - Ospedale Civile - Sc Cardiologia Area Nord, Guastalla, RE
  - Arcispedale Santa Maria Nuova - S.C. Cardiologia, Reggio Emilia, RE
  - Ospedale Giovanni Paolo Ii - U.O.C. Cardiologia-Utic, Ragusa, RG
  - Nuovo Ospedale Dei Castelli - U.O.C. Di Cardiologia E Utic, Ariccia, RM
  - Campus Biomedico - Cardiologia, Roma, RM
  - P.O. San Filippo Neri - Asl Roma 1 - Uoc Cardiologia E Utic, Roma, RM
  - Ospedale San Camillo - Uosd Servizi Cardiologici Integrati, Roma, RM
  - Ifo- Istituto Naz. Tumori Regina Elena - Uo Cardiologia, Roma, RM
  - Policlinico Agostino Gemelli - Uo Cardiologia Per Sc E Riab. Cardiolog., Roma, RM
  - Ospedale G. Ceccarini - Cardiologia-Utic, Riccione, RN
  - Aou S. Giovanni Di Dio-Ruggi D'Aragona - Cardiologia Intensiva, Salerno, SA
  - Ospedale Dell'Alta Val D'Elsa - Uosd Cardiologia-Utic, Poggibonsi, SI
  - Ospedale San Bartolomeo - U.O. Cardiologia Clinica-Riabilitativa, Sarzana, SP
  - Ospedale E. Muscatello - U.O. Di Cardiologia - Utic, Augusta, SR
  - Ospedale Di Castellaneta - S.C. Cardiologia, Castellaneta, TA
  - Ospedale Civile M. Giannuzzi - Cardiologia E Utic, Manduria, TA
  - Presidio Ospedaliero Della Valle D'Itria - Struttura Complessa Di Cardiologia, Martina Franca, TA
  - Ospedale Civile G. Mazzini - Cardiologia Utic Ed Emodinamica, Teramo, TE
  - Ospedale Santa Maria Del Carmine - Cardiologia, Rovereto, TN
  - Ospedale San Luigi Gonzaga - S.C.D.O. Cardiologia, Orbassano, TO
  - Ospedale Civile E. Agnelli - Sc Di Cardiologia, Pinerolo, TO
  - Ospedale Degli Infermi, Sc Cardiologia, Rivoli, TO
  - Aou Citta' Della Salute E Della Scienza - S.C.D.U. Cardiologia, Torino, TO
  - Ospedale Mauriziano Umberto I - Sc Cardiologia, Torino, TO
  - Ospedale Humanitas Gradenigo - Cardiologia, Torino, TO
  - Ospedale Giovanni Bosco - Sc Cardiologia, Torino, TO
  - Ospedale Ss. Vito E Spirito - U.O.S. Di Cardiologia, Alcamo, TP
  - Azienda Ospedaliera Santa Maria - S.C. Di Cardiologia, Terni, TR
  - Asui Trieste - S.C. Centro Cardiovascolare, Trieste, TS
  - Pou Santa Maria Della Misericordia - S.O.C. Cardiologia, Udine, UD
  - Presidio Ospedaliero Di Saronno - U.O.C. Di Cardiologia, Saronno, VA
  - Ospedale Civile - U.O. Cardiologia, Mirano, VE
  - Ospedale Civile - U.O.C. Cardiologia, Arzignano, VI
  - Ospedale Sacro Cuore - U.O. Di Cardiologia, Negrar, VR
  - Ospedale Miulli - U.O.C. Cardiologia - Utic, Acquaviva delle Fonti
  - Ospedale Ss. Trinita' - S.C. Di Cardiologia, Borgomanero
  - Az. Ospedaliera S. Anna E S. Sebastiano - Uoc Medicina E Chirurgia D'Urgenza, Caserta
  - Ospedale Policlinico Ss. Annunziata - Medicina Generale Ii, Chieti
  - Arcispedale Sant'Anna - U.O. Cardiologia - Utic, Ferrara
  - Ospedale Generale Di Zona - U.O. Cardiologia - Utic, Giugliano in Campania
  - Fondazione Pascale - S.C. Cardiologia, Napoli
  - Ospedale San Gennaro - U.O. Cardiologia E Riabilitazione Card., Napoli
  - Aou Maggiore Della Carita' - Cardiologia Ii, Novara
  - Ospedale Ss. Cosma E Damiano - U. O. Cardiologia - Utic, Pescia
  - Ospedale Santa Maria Delle Grazie - U.O. Cardiologia - Utic, Pozzuoli
  - Ospedale Sandro Pertini, Uoc Cardiologia, Roma
- Netherlands (8):
  - Jeroen Bosch Ziekenhuis - Research Cardiologie, 's-Hertogenbosch
  - Rijnstate Ziekenhuis - Afdeling Cardioresearch, Arnhem
  - Tergooi - Poli cardiologie / poli 2, Blaricum
  - Amphia Ziekenhuis - Research Cardiologie, Breda
  - Martini Ziekenhuis - Dept. Cardio Research Noord BV, Groningen
  - Diakonessenhuis - Research Cardiologie, Utrecht
  - University Medical Center Utrecht - Cardiologie, Utrecht
  - Máxima Medisch Centrum - Poli Cardiologie, Veldhoven
- Portugal (5):
  - Prof. Doutor Fernando Fonseca EPE Hospital, Cardiologia, Amadora
  - Hospital Nossa Senhora do Rosário, Cardiology, Barreiro
  - Hospital da Luz, Lisbon
  - Hospital de Santa Cruz, Cardiology, Lisbon
  - Hospital Santa Maria, Cardiology, Lisbon
- Spain (19):
  - Hospital del Mar (Parc de Salut Mar),Cardiologa I Unitat Coronaria, Barcelona
  - Hospital Médico-Quirúrgico, Cardiology, Jaén
  - Clínica Anderson, Oncología Médica, Madrid
  - Clínica Medicentro, Cardiología, Madrid
  - Hopsital Puerta de Hierro, Madrid
  - Hospital La Moraleja, Servicio de Cardiología, Madrid
  - Hospital La Paz, Madrid
  - Hospital La Zarzuela, Madrid
  - Hospital Montepríncipe, Cardiología, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Rúber Internacional, Oncología, Madrid
  - Hospital Universitario Gregorio Marañón, Servicio de Cardiología, Madrid
  - Hospital Virgen de Arrixaca - Cardiologia, Murcia
  - Hospital de Salamanca, Cardiología, Salamanca
  - Hospital Universitario Virgen Macarena, Cardiologia, Seville
  - Hospital de Torrejón, Torrejón de Ardoz
  - Hospital Universitario Río Hortega, Cardiología, Valladolid
  - University Clinical Hosp. de Valladolid, Cardiología, Valladolid
  - Hospital Clínico "Lozano Blesa", Cardiologia, Zaragoza

REFERENCES:
- [Derived] Gulizia MM, Turazza FM, Ameri P, Alings M, Collins R, De Luca L, Di Nisio M, Lucci D, Gabrielli D, Janssens S, Parrini I, Pinto FJ, Zamorano J, Colivicchi F; BLITZ-AF Cancer Investigators. Characteristics and Management of Patients With Cancer and Atrial Fibrillation: The BLITZ-AF Cancer Registry. JACC Adv. 2024 May 24;3(7):100991. doi: 10.1016/j.jacadv.2024.100991. eCollection 2024 Jul. PMID 39130025